CLINICAL TRIAL: NCT02606630
Title: A [C-11]-PBR28 Positron Emission Tomography Study to Evaluate the Effect of ABT-555 on Central Nervous System Inflammation in Subjects With Relapsing Forms of Multiple Sclerosis
Brief Title: [11C]-PBR28 Positron Emission Tomography Study to Evaluate the Effect of ABT 555 in Subjects With Relapsing Forms of Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-561; 2015-001176-22 (EudraCT Number)
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — elezanumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-555 (Experimental): ABT-555 will be administered at Visit 4 for Part 2 only
  Interventions: Drug: ABT-555

INTERVENTIONS:
Drug: ABT-555 — ABT-555 will be administered on Visit 4 in Part 2 only

SUMMARY:
This open-label positron emission tomography (PET) study is designed to determine the effect of ABT-555 on translocator protein expression level in participants with relapsing forms of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of relapsing-remitting MS (RRMS) or relapsing secondary progressive MS (SPMS)

Neurologically stable at Screening, in the investigator's judgment and not actively experiencing or recovering from a recent relapse in the 30 days preceding the Screening Visit

A Kurtzke Expanded Disability Status Scale (EDSS) score of 1.0 to 6.0, inclusive at the Screening Visit

High or mixed affinity binder of the TSPO, as determined by rs6971 polymorphism genotyping at screening

Exclusion Criteria:

Diagnosis of primary progressive or non-relapsing secondary progressive MS

Smoking more than 10 cigarettes per day or use of a nicotine patch

Known history of, or positive screening test result for hepatitis C virus or hepatitis B virus

Varicella or herpes zoster virus infection or any severe viral infection within 6 weeks before Screening

Any type of live virus vaccine from 4 weeks before randomization

History of abnormal laboratory results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in translocator protein expression | Day 0 and 109 days
  Compare 2 dynamic positron emission tomography scans to examine the effect of a single administration of ABT-555 on translocator protein expression

CONTACTS AND LOCATIONS:
Overall Officials: Steven Greenberg, MD, Study Director — AbbVie
Locations (2):
- United Kingdom (2):
  - Site Reference ID/Investigator# 141463, London
  - Site Reference ID/Investigator# 141461, Whitechapel